CLINICAL TRIAL: NCT00836589
Title: GALAXY Registry: Long-term Evaluation of the Linox Family ICD Leads Registry
Brief Title: Long-term Evaluation of the Linox Family ICD Leads Registry (GALAXY)
Acronym: GALAXY
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GALAXY
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Patients Indicated for an ICD
Keywords: Long-term safety and reliability of ICD leads

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data Collection Group
  Interventions: Device: ICD Therapy - ICD Lead Registry

INTERVENTIONS:
Device: ICD Therapy - ICD Lead Registry — Collecting long-term safety and efficacy data on a family of market-released ICD leads.

SUMMARY:
The objective of this study is to confirm the long-term safety and reliability of the Linox Lead System as used with BIOTRONIK ICDs. The GALAXY registry will provide data to fully characterize ICD lead failures, from implant through 5 years, including those failures contributing to patients losing pacing or defibrillation therapy.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, non-randomized, 5-year data collection registry. Eligible patients must have been successfully implanted with a Linox Lead System connected to a BIOTRONIK ICD and consented and enrolled between 1-45 days following implant. This study is designed to be a post-implant (office-based) registry, and patients are meant to be seen according to each institution's standard of care, but not to exceed a follow-up time frame of every 6 months. At least 2000 patients will be enrolled in this registry, and each patient will be followed for five years post-implant.

Safety will be evaluated based on the analysis of the overall incidence of lead-related adverse events that require additional invasive intervention to resolve. In addition, each individual adverse event will be separately investigated. Lead parameters for sensing, pacing thresholds, and impedance will also be evaluated. An independent Clinical Events Committee will review and adjudicate all adverse events that occur during the study according to the protocol definitions.

ELIGIBILITY:
Inclusion Criteria:

* Successfully implanted Linox Lead System connected to a BIOTRONIK ICD, from 1-45 days prior to enrollment
* Able to understand the nature of the registry and provide informed consent
* Available for follow-up visits on a regular basis at the investigational site
* Age greater than or equal to 18 years

Exclusion Criteria:

* Enrolled in any IDE clinical study
* Planned cardiac surgical procedures or investigational measures within the next 6 months
* Expected to receive a heart transplant within 1 year
* Life expectancy less than 1 year
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Pregnancy
* Inability to provide date of implant, devices implanted, age, gender, and whether the patient experienced any protocol-defined adverse events since implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be obtained from the investigators' general patient population according to the inclusion and exclusion criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 1997 (Actual)
Dates: Start 2008-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (85):
  - Albertville, Alabama
  - Birmingham, Alabama
  - Gadsden, Alabama
  - Jasper, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Burbank, California
  - Fairfield, California
  - Fountain Valley, California
  - Glendale, California
  - Hawthorne, California
  - Inglewood, California
  - Los Angeles, California
  - Mission Viejo, California
  - Northridge, California
  - Rancho Mirage, California
  - Santa Barbara, California
  - Santa Maria, California
  - Torrance, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Brooksville, Florida
  - Daytona Beach, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - Pensacola, Florida
  - Port Charlotte, Florida
  - Atlanta, Georgia
  - Alton, Illinois
  - Centralia, Illinois
  - Chicago, Illinois
  - Hammond, Indiana
  - Jeffersonville, Indiana
  - Owensboro, Kentucky
  - Lafayette, Louisiana
  - Lake Charles, Louisiana
  - Marrero, Louisiana
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Rockville, Maryland
  - Salisbury, Maryland
  - Grand Rapids, Michigan
  - Ypsilanti, Michigan
  - Biloxi, Mississippi
  - Bridgeton, Missouri
  - Crystal City, Missouri
  - St Louis, Missouri
  - Haddon Heights, New Jersey
  - Rochester, New York
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Gastonia, North Carolina
  - Greensboro, North Carolina
  - Grand Forks, North Dakota
  - Columbus, Ohio
  - Massillon, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Salem, Oregon
  - Tualatin, Oregon
  - Chinchilla, Pennsylvania
  - Phoenixville, Pennsylvania
  - Yardley, Pennsylvania
  - Columbia, South Carolina
  - Florence, South Carolina
  - Greenville, South Carolina
  - Greenwood, South Carolina
  - Lancaster, South Carolina
  - Rock Hill, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Kingwood, Texas
  - McAllen, Texas
  - McKinney, Texas
  - Yakima, Washington

REFERENCES:
- [Derived] Good ED, Cakulev I, Orlov MV, Hirsh D, Simeles J, Mohr K, Moll P, Bloom H. Long-Term Evaluation of Biotronik Linox and Linox(smart) Implantable Cardioverter Defibrillator Leads. J Cardiovasc Electrophysiol. 2016 Jun;27(6):735-42. doi: 10.1111/jce.12971. Epub 2016 May 3. PMID 26990515

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Data Collection Group
Started | 1997
Completed | 731
Not Completed | 1266
Not completed — Lost to Follow-up | 246
Not completed — Death | 429
Not completed — Withdrawal by Subject or Physician | 591

BASELINE CHARACTERISTICS:
Arm/Group | Data Collection Group
Number analyzed (Participants) | 1997
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Enrollment | 64.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 537
  Male | 1460
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1298
  Race: Black or African American | 288
  Race: Hispanic or Latino | 244
  Race: Unknown | 139
  Race: Asian | 21
  Race: Native Hawaiian or Other Pacific Islander | 4
  Race: Amerian Indian or Alaska Native | 3
Height [Mean (Standard Deviation); unit: in] | 68.0 (4.0)
Weight [Mean (Standard Deviation); unit: lbs] | 194.2 (49.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are Free of Complications Related to the Linox ICD Lead
Description: The overall incidence of complications (serious adverse events that require additional invasive intervention to resolve or specific non-invasive actions) related to the Linox ICD leads implanted with a market-released BIOTRONIK ICD device was evaluated. This was evaluated as a serious adverse event free-rate (SAEFR).
Time Frame: 5 years
Population: The evaluable subject population is the sum of the total unique subjects who completed the 5-year follow-up and/or who experienced a primary endpoint adverse event.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Data Collection Group
Number analyzed (Participants) | 777
percentage of subjects | 90.9 [88.6 to 92.8]
Statistical Analysis 1: Comparison: Data Collection Group; Test type: Non-Inferiority — Estimated SAEFR at 5 years is 92.5% with a 5% non-inferiority margin (87.5%). Type I error (alpha) is 0.05 (one-sided for non-inferiority). Statistical power is 80%; p = 0.0020, Binomial Proportion

2. Primary Outcome: Number of Subjects Who Experienced Primary Outcome 1 Complication(s) Per Individual Complication Type
Description: Evaluation of the individual types of serious adverse events (SAEs) contributing to primary outcome 1 and their associated SAE category.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Data Collection Group
Number analyzed (Participants) | 777
Participants
  Low lead impedance, potential insulation breach | 25
  High lead impedance, potential conductor fracture | 20
  Lead noise or oversensing | 17
  Lead dislodgement (>180 days post-implant) | 6
  Lead undersensing or loss of sensing | 2
  Inability to defibrillate or pace | 1
  No slack in lead due to probable dislodgement | 1
  Noise consistent with probable fracture | 1
  Tension pneumothorax | 1

3. Secondary Outcome: Number of Subjects Who Experienced Serious Adverse Event(s) Excluded From Primary Outcome 1 (ICD, Device, and Implant Procedure Related) Through 5 Years Post-Implant.
Time Frame: 5 years
Population: The evaluable subject population is the sum of the total unique subjects who completed the 5-year follow-up and/or who experienced a secondary endpoint adverse event (ICD lead, device, implant procedure, or other related).
Measure: Count of Participants; unit: Participants
Arm/Group | Data Collection Group
Number analyzed (Participants) | 830
Participants
  Total related to the ICD lead | 42
  Total device related | 6
  Total implant procedure related | 58
  Total other AEs | 22

4. Secondary Outcome: Number of Subjects Who Experienced Serious Adverse Event(s) Excluded From Primary Outcome 1 (RA Lead Related) Through 5 Years Post-Implant.
Time Frame: 5 years
Population: The evaluable subject population is the sum of the total unique subjects who completed the 5-year follow-up and had an RA lead implanted for any duration and/or who experienced a secondary endpoint adverse event (RA lead related).
Measure: Number; unit: subjects with adverse event
Arm/Group | Data Collection Group
Number analyzed (Participants) | 562
subjects with adverse event | 39

5. Secondary Outcome: Pacing Threshold Measurements for the Linox Lead System at Scheduled GALAXY Registry Follow-ups Through 5 Years Post-implant.
Description: Pacing thresholds performed at 0.5 ms pulse-width were requested. Threshold data reported below was collected at 0.5 ms pulse-width. The mean pacing threshold is calculated as a mean across all study visits.
Time Frame: 5 years
Population: 17 subjects were excluded due to incomplete data.
Measure: Mean (Standard Deviation); unit: Volts (V)
Groups:
- Linox Lead System: Linox leads including S, SD, T, and TD models, Linox smart leads including smart S, smart SD, and smart TD models.
Arm/Group | Linox Lead System
Number analyzed (Participants) | 1980
Volts (V) | 0.64 (0.35)

6. Secondary Outcome: Sensing Measurements for the Linox Lead System at Scheduled GALAXY Registry Follow-ups Through 5 Years Post-implant.
Description: The mean sensing measurement is calculated as a mean across all study visits.
Time Frame: 5 years
Population: 17 subjects were excluded due to incomplete data.
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Linox Lead System
Number analyzed (Participants) | 1980
millivolts (mV) | 12.77 (5.40)

7. Secondary Outcome: Pacing Impedance Measurements for the Linox Lead System at Scheduled GALAXY Registry Follow-ups Through 5 Years Post-implant.
Description: The mean pacing impedance measurement is calculated as a mean across all study visits.
Time Frame: 5 years
Population: 17 subjects were excluded due to incomplete data.
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Linox Lead System
Number analyzed (Participants) | 1980
ohms | 552.9 (136.4)

8. Secondary Outcome: Individual Electrical Parameters (Pacing Threshold) of Each Linox Lead System Model.
Description: Pacing thresholds performed at 0.5 ms pulse-width were requested. Threshold data reported below was collected at 0.5 ms pulse-width. The mean pacing threshold of each Linox Lead System model was calculated as a mean across all study visits.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: Volts (V)
Arm/Group | Linox S | Linox SD | Linox T | Linox TD | Linox Smart S | Linox Smart SD | Linox Smart TD
Number analyzed (Participants) | 338 | 1352 | 1 | 88 | 24 | 173 | 4
Volts (V) | 0.62 (0.31) | 0.64 (0.33) | 0.50 (0.00) | 0.76 (0.62) | 0.59 (0.22) | 0.66 (0.46) | 0.67 (0.31)

9. Secondary Outcome: Individual Electrical Parameters (Sensing) of Each Linox Lead System Model.
Description: The mean sensing measurements of each Linox Lead System model were calculated as a mean across all study visits.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Linox S | Linox SD | Linox T | Linox TD | Linox Smart S | Linox Smart SD | Linox Smart TD
Number analyzed (Participants) | 338 | 1352 | 1 | 88 | 24 | 173 | 4
millivolts (mV) | 13.66 (5.69) | 12.71 (5.41) | 5.63 (0.81) | 10.96 (4.06) | 13.12 (5.14) | 12.25 (4.93) | 10.25 (1.46)

10. Secondary Outcome: Individual Electrical Parameters (Pacing Impedance) of Each Linox Lead System Model.
Description: The mean pacing impedance of each Linox Lead System model was calculated as a mean across all study visits.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Linox S | Linox SD | Linox T | Linox TD | Linox Smart S | Linox Smart SD | Linox Smart TD
Number analyzed (Participants) | 338 | 1352 | 1 | 88 | 24 | 173 | 4
ohms | 550.9 (105.3) | 541.8 (120.5) | 812.0 (202.5) | 784.8 (306.2) | 541.5 (106.5) | 546.0 (99.2) | 734.4 (253.8)

ADVERSE EVENTS:
Time Frame: Implant to Study Exit (up to 5 years)
Arm/Group | Data Collection Group
All-Cause Mortality (participants affected / at risk) | 429/1997
Serious Adverse Events (participants affected / at risk) | 215/1997
Other Adverse Events (participants affected / at risk) | 31/1997
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Data Collection Group (N=1997)
ICD lead dislodgement (occuring <= 180 days post-implant procedure) (Cardiac disorders) | 24 (25)
ICD lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 12 (13)
ICD lead related cardiac perforation with or without tamponade (Cardiac disorders) | 5 (6)
ICD lead impedance out of range, low impedance, potential insulation break (Cardiac disorders) | 25 (25)
ICD lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 18 (18)
Other ICD lead related: lead noise or oversensing (Cardiac disorders) | 17 (17)
ICD lead dislodgement (occuring > 180 days post-implant procedure) (Cardiac disorders) | 6 (6)
ICD lead undersensing or loss of sensing (Cardiac disorders) | 2 (2)
ICD lead inability to defibrillate or pace (Cardiac disorders) | 1 (1)
Other ICD lead related: no slack in the lead due to probable dislodgement (Cardiac disorders) | 1 (1)
Other ICD lead related: noise consistent with probable fracture (Cardiac disorders) | 1 (1)
Other ICD lead related: tension pneumothorax (Cardiac disorders) | 1 (1)
Pocket pain (Cardiac disorders) | 2 (2)
Unable to interrogate device (Cardiac disorders) | 2 (2)
Suspected generator failure (Cardiac disorders) | 1 (1)
Premature battery depletion, warranting device replacement (Cardiac disorders) | 1 (1)
RA lead dislodgement (Cardiac disorders) | 18 (18)
RA lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 2 (3)
RA lead undersensing or loss of sensing (Cardiac disorders) | 3 (3)
RA lead oversensing or noise (Cardiac disorders) | 1 (1)
RA lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 1 (1)
RA lead loose set screw (Cardiac disorders) | 1 (1)
Infection not due to secondary infection (Infections and infestations) | 27 (27)
Hematoma (Surgical and medical procedures) | 7 (7)
Loose set screw (Surgical and medical procedures) | 4 (4)
Non-healing pocket dehiscence requiring intervention (Surgical and medical procedures) | 3 (3)
Bleeding (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Surgical and medical procedures) | 1 (1)
Impending erosion (Surgical and medical procedures) | 1 (1)
Pain at insertion site (Surgical and medical procedures) | 1 (1)
Pocket erosion (Surgical and medical procedures) | 1 (1)
Pulmonary embolism (unrelated to ICD lead) (Surgical and medical procedures) | 1 (1)
Shock coils reversed in header (Surgical and medical procedures) | 1 (1)
Infection due to secondary infection (Infections and infestations) | 14 (14)
Twiddler's syndrome (General disorders) | 5 (6)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Pulseless electrical activity (PEA) arrest (Cardiac disorders) | 1 (1)
LV lead dislodgement (Cardiac disorders) | 1 (1)
Thrombus attached to ICD lead (unrelated to ICD lead) (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Data Collection Group (N=1997)
ICD lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 2 (2)
ICD lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 2 (2)
RA lead dislodgement (Cardiac disorders) | 11 (11)
RA lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 1 (1)
RA lead oversensing or noise (Cardiac disorders) | 2 (2)
Infection not due to secondary infection (Infections and infestations) | 1 (1)
Hematoma (Surgical and medical procedures) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agree to submit copies of any manuscript proposed for publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may extend such review period for another 90 days to file patent applications or take other steps to protect its intellectual property interests, or to remove from the paper or presentation any language that is detrimental to Sponsor's intellectual property interests